CLINICAL TRIAL: NCT06551311
Title: To Explore Efficacy and Load of Eccentric Cycling Training in Older CKD Patients with or Without Sarcopenia
Brief Title: The Effects of Eccentric Cycling Exercise Program in Chronic Kidney Disease Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Kun-Ling Tsai, Professor and Chair Department of Physical Therapy/Institute of Allied Health Science National Cheng Kung University, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A-BR-110-109
Record Dates: First submitted 2024-07-16; First posted 2024-08-13 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Chronic Kidney Disease
Keywords: Eccentric Cycling Exercise Training; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: In this randomized controlled trial, participants were assigned to one of three groups: the concentric cycling exercise training group, the eccentric cycling exercise training group, or the control group with no exercise intervention. Over eight weeks, participants completed 24 exercise sessions, three times per week, with each session lasting between 20 and 30 minutes. The allocation of participants to groups was determined using a random numbers table.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (No Intervention): Receive regular health care
- The concentric cycling exercise training group (Experimental): Over eight weeks, participants completed 24 exercise sessions, three times per week, with each session lasting between 20 and 30 minutes under concentric cycling exercise training.
  Interventions: Behavioral: cycling training exercise
- The eccentric cycling exercise training group (Experimental): Over eight weeks, participants completed 24 exercise sessions, three times per week, with each session lasting between 20 and 30 minutes under eccentric cycling exercise training.
  Interventions: Behavioral: cycling training exercise

INTERVENTIONS:
Behavioral: cycling training exercise — Participants were randomly allocated to one of three groups: control (CTL), concentric cycling training (CON), or eccentric cycling training (ECC).
  CTL: Received standard health education guidance.
  CON and ECC: Participants in both the CON and ECC groups engaged in 24 exercise sessions, performed three times per week, lasting between 20 and 30 minutes. Both groups trained on a stationary bicycle, with the CON group performing concentric cycling and the ECC group performing eccentric cycling. The exercise intensity for both groups was set to a rating of perceived exertion (RPE) level of 13. Sessions began at 20 minutes and increased incrementally by 3-5 minutes each week until participants could sustain a 30-minute duration. The initial exercise intensity was set at 50% of the maximal output determined by a cardiopulmonary exercise test, and it was progressively increased by 5-10% of the estimated target power weekly, with adjustments made primarily to maintain an RPE of 13.
  Arms: The concentric cycling exercise training group; The eccentric cycling exercise training group

SUMMARY:
Progress in medical technology, enhancements in environmental cleanliness, and elevated living conditions have notably prolonged the mean life expectancy, resulting in a swift increase in the aging population. The prevalence of Chronic Kidney Disease (CKD) is more pronounced among the elderly in contrast to younger demographics. With the aging of the CKD population, the capacity to autonomously handle daily activities becomes a critical concern. This demographic frequently encounters concurrent health conditions, a decrease in self-care capabilities, general health decline, and diminished quality of life.

Recent studies suggest that physical activity has the potential to enhance cardiovascular health, cardiopulmonary endurance, muscle strength, quality of life, uremic toxin management, and inflammation levels among individuals with CKD. Given that CKD patients often exhibit sedentary behavior and reduced exercise capacity, eccentric cycling exercises may be particularly well-suited for this demographic.

Compared to concentric contractions, eccentric contractions subject the muscles to higher tension. Since muscle growth partially depends on the "stress exerted on muscle fibers"-meaning the greater the stress, the more stimulation the muscles receive-training focused on eccentric contractions could provide more stimulation and promote greater muscle growth.

In recent studies, eccentric cycling has emerged as a feasible and promising aerobic exercise intervention. It can provide a safe and appropriate amount of exercise while relatively reducing joint pressure. This novel combined aerobic and anaerobic exercise method is particularly beneficial for individuals with weaker lower limb muscles, lower joint pressure tolerance, poor metabolic and cardiovascular function, and a tendency to fatigue.

DETAILED DESCRIPTION:
The previous study did not examine the impact of eccentric cycling exercise training on individuals with CKD. This study focuses on exploring the effects of eccentric cycling exercise on various aspects including body composition, functional capacity, flexibility, muscle strength, exercise capacity, pulmonary function, quality of life, and renal function in CKD patients. A comparison will be made between eccentric cycling exercise training, concentric cycling exercise training, and the usual care provided. The goal is to provide a clearer understanding of how eccentric cycling exercise can benefit individuals with CKD.

ELIGIBILITY:
This study will be conducted in collaboration with the Departments of Nephrology and Geriatric Medicine at National Cheng Kung University Hospital, Taiwan. Participants will be recruited as voluntary subjects from outpatient clinics. The attending physician will assess eligible patients. After the study's purpose and methodology are explained by the research staff and patients consent to participate, block randomization will be used to assign participants into one of three groups randomly. The allocation results will be securely stored by the principal investigator.

Inclusion Criteria:

* (1) Clinical diagnosis of CKD
* (2) eGFR <60 ml/min/1.73m^2 or undergoing routine dialysis
* (3) Must be able to communicate normally, understand and comply with instructions.
* (4) Must be able to walk independently.

Exclusion Criteria:

* (1) Clinical diagnosis of acute renal failure
* (2) Hospitalization for acute illness within the past three months
* (3) Clinical diagnosis of severe joint disease and lower extremity surgery
* (4) Clinical diagnosis of severe neurological disease
* (5) Clinical diagnosis of severe cardiovascular disease
* (6) Unconsciousness or lack of ability to cooperate with the assessment

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary Exercise Testing (CPET) | at Baseline, midterm test (at 4 weeks), post-test (at 8 weeks), and follow-up test (at 12 weeks)
  CPET evaluates both submaximal and peak exercise responses of the pulmonary, cardiovascular, hematopoietic, neuropsychological, and skeletal muscle systems for diagnostic and prognostic assessment. It aims to assess exercise performance, functional capacity, and impairment by identifying undiagnosed exercise intolerance and symptoms.
Pulmonary function test | at Baseline, midterm test (at 4 weeks), post-test (at 8 weeks), and follow-up test (at 12 weeks)
  Spirometry is a physiological test that measures the ability to inhale and exhale air over time. The main spirometry results are forced vital capacity (FVC), forced expiratory volume in the first second (FEV1), and the FEV1/FVC ratio.
Maximum respiratory pressure (MIP/MEP) | at Baseline, midterm test (at 4 weeks), post-test (at 8 weeks), and follow-up test (at 12 weeks)
  Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) measurements help evaluate respiratory muscle weakness.
Six Minute Walk Test (6MWT) | at Baseline, midterm test (at 4 weeks), post-test (at 8 weeks), and follow-up test (at 12 weeks)
  The American Thoracic Society developed the 6-minute walk test (6MWT) to assess patients with cardiopulmonary issues and has since been used for various other conditions. It is a low-intensity, submaximal exercise test that measures aerobic capacity, endurance, and oxygen saturation.
Lower limb strength-Knee Extension Strength Test | at Baseline, midterm test (at 4 weeks), post-test (at 8 weeks), and follow-up test (at 12 weeks)
  The Knee Extension Strength Test is a clinical assessment used to measure the maximal force production of the quadriceps muscles in both legs (bilateral lower limb strength). It's a valuable tool for identifying muscle weakness, tracking progress after injury or rehabilitation, and guiding treatment decisions.

SECONDARY OUTCOMES:
Physical fitness-Body composition | at Baseline, midterm test (at 4 weeks), post-test (at 8 weeks), and follow-up test (at 12 weeks)
  Body composition is a key component for maintaining good general. Body composition refers to the distribution of fat, muscle, bone, and other tissues that make up your body. It is often expressed as the percentage of total body weight that consists of fat and/or lean body mass. Body composition offers numerous insights into health, fitness, and nutritional status.
  Utilize Bioelectrical Impedance Analysis (BIA) equipment to assess a range of body composition parameters, including high (m^2), weight (kg), body fat (%), Skeletal muscle rate (%), basal metabolic rate, and BMI (kg/m^2).
Physical fitness-Flexibility | at Baseline, midterm test (at 4 weeks), post-test (at 8 weeks), and follow-up test (at 12 weeks)
  Flexibility, the ability to move joints through their full range of motion, is key for physical health. Upper limb test: Apley scratch test assess shoulder flexibility, helping gauge overall mobility.
Physical fitness-muscle strength | at Baseline, midterm test (at 4 weeks), post-test (at 8 weeks), and follow-up test (at 12 weeks)
  Muscle strength is characterized as the maximum force that a muscle or a group of muscles can produce at a specific or predetermined velocity. In essence, it refers to the capacity of skeletal muscle to generate force, which is crucial for ensuring stability and mobility within the musculoskeletal system.
  Upper arm testing-hand grip test: The purpose of the handgrip strength test is to measure the maximum isometric strength of the hand and forearm muscles. The subject holds the dynamometer in the hand to be tested, with the arm at right angles and the elbow by the side of the body. The handle of the dynamometer is adjusted if required - the base should rest on the first metacarpal (heel of palm), while the handle should rest on middle of the four fingers. When ready the subject squeezes the dynamometer with maximum isometric effort, which is maintained for about 5 seconds. No other body movement is allowed. The subject should be strongly encouraged to give a maximum effort.
  Lower
Quality of life indicators-SF-36 Questionnaire | at Baseline and follow up test (at 12 weeks)
  SF-36 is a very popular instrument for evaluating Health-Related Quality of Life.
  The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). the score is in two steps. Precoded numerical values are first recorded by the scoring key in eight scales. Each item is rated, and a higher number indicates that the subject is in better overall health. Also, each item is graded on a scale of 0 to 100, with 0 and 100 as the lowest and highest possible scores. The eight scale scores are produced in step 2 by averaging the items on the same scale.
  There are two distinct concepts measured by the SF-36: a physical dimension, represented by the Physical Component Summary (PCS), and a mental dimension, represented by the Mental Component Summary (MCS). All scales contribute in different proportions to the scoring of both PCS and MCS measures.
Quality of life indicators- KDQOL Questionnaire | at Baseline and follow up test (at 12 weeks)
  Health-related quality of life is a crucial outcome for the chronic kidney disease population, the Kidney Disease Quality of Life (KDQOL) questionnaire is commonly used as an integral part of clinical evaluations. The KDQOL-36™ is a short form that includes the SF-12 as generic core plus the burden of kidney disease, symptoms/problems of kidney disease, and effects of kidney disease scales from the KDQOL-SF™v1.3.
  Items 1-12: SF-12 Items 13-16: Burden of kidney disease Items 17-28: Symptoms/problems Items 29-36: Effects of kidney disease

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hostipal, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD sharing plan will be decided after summarized data being published.